CLINICAL TRIAL: NCT07039851
Title: Creative Drama and Gamification-Based Educational Experience: Its Effect on Children's Nature Connectedness and Recycling Behaviors
Brief Title: CreativeDrama and GamificationBased
Acronym: Creative Drama
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Merve Kolcu, Assistant professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025/06
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Creative Drama; Gamification
Keywords: Creative drama; Gamification; Nature connectedness; Recycling behaviors; Environmental education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Creative drama and gamification sessions will be conducted under the guidance of a creative drama facilitator and will consist of four stages:
  Warm-up phase (10 minutes)
  Games and activities phase (30 minutes)
  Improvisation and creative participation phase (30 minutes)
  Evaluation and feedback phase (20 minutes)
  In each session, students will be divided into different groups of equal size to promote cooperation and interaction.
  The experimental group will receive training based on creative drama and gamification, while the control group will be taught using traditional instructional methods. Both groups will participate in two sessions, held once a week.
  The content of the training will be structured around the themes of nature connectedness and recycling behaviors, with each session lasting approximately 90 minutes.
  Interventions: Other: Experimental
- No Intervention (No Intervention): The control group will be taught the same topics using a traditional instructional method, without the use of creative drama or gamification elements.

INTERVENTIONS:
Other: Experimental — Each session in the experimental group includes four phases:
  1. Warm-up (10 min): Students engage in ice-breakers and movement activities to relax and prepare mentally and physically.
  2. Games & Activities (30 min): Drama and game-based tasks related to nature and recycling promote experiential learning and teamwork.
  3. Improvisation (30 min): Students take part in role-plays and skits (e.g., acting as a tree or a recycled item) to build empathy and deepen their connection to environmental themes.
  4. Evaluation (20 min): Students reflect on their learning, share feelings, and receive feedback. Facilitators summarize key points and reinforce the session's goals.
  Arms: Experimental

SUMMARY:
The aim of this study is to examine the effect of a creative drama and gamification-based educational experience on children's levels of nature connectedness and recycling behaviors. With the increasing environmental problems today, instilling environmental awareness in children at an early age and helping them establish a bond with nature is of great importance for a sustainable future. In this context, creative drama stands out as an effective method in shaping environmental attitudes, as it supports children's emotional development and enhances their ability to empathize. Gamification, on the other hand, is a pedagogical strategy that increases children's active participation in learning processes and boosts their motivation.

In the study, an experimental design will be used, and a group of students will participate in an educational program themed around nature and recycling, incorporating creative drama and gamification activities. At the end of the program, children's nature connectedness and recycling behaviors will be measured, and pre-test-post-test comparisons will be made. Nature connectedness is defined as an individual's perception of nature as a whole and seeing themselves as a part of that whole, and it is strongly associated with environmentally friendly behaviors. Recycling behaviors include individuals' voluntary efforts to separate and repurpose waste.

This study aims to reveal how creative and interactive learning methods influence children's environmental awareness and behaviors, and it seeks to contribute to the development of environmental education programs.

DETAILED DESCRIPTION:
Research Design This study will be conducted using a quantitative research method within a randomized controlled experimental design, employing a pre-test and post-test approach.

Population and Sample The study population consists of students enrolled in the 5th and 6th grades of middle schools affiliated with the Istanbul Provincial Directorate of National Education. The experimental group will receive an educational program based on creative drama and gamification, while the control group will not receive any intervention during this period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female students aged 10 to 12 years.

Enrolled in 5th or 6th grade at middle schools affiliated with the Istanbul Provincial Directorate of National Education.

Voluntary participation with parental consent.

Able to attend all sessions and actively participate in the educational activities.

Exclusion Criteria:

-

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Nature Connectedness Scale | 5 minutes
  In this study, the Nature Connectedness Scale developed by Cheng and Monroe (2012) and adapted into Turkish by Alkış Küçükaydın (2024) will be used to measure children's emotional and cognitive levels of connectedness to nature. The scale consists of 16 items designed to assess children's relationships with nature across emotional, empathic, and responsibility dimensions.
  The instrument uses a five-point Likert scale: "Strongly Disagree", "Disagree", "Neutral", "Agree", and "Strongly Agree."
The Recycling Scale for Middle School Students | 5 minutes
  The Recycling Scale for Middle School Students consists of a structure with 15 items grouped under three factors. However, one item was removed from the scale due to its standardized regression weight falling below 0.5, and Confirmatory Factor Analysis (CFA) was conducted again. As a result, the final version of the scale was confirmed to include 14 items under three dimensions: awareness, behavior, and attitude. The reliability of the scale was determined using Cronbach's Alpha, yielding a value of 0.856, indicating high internal consistency.
Demographic Information Form | 5 minutes
  The Demographic Information Form developed by the researcher will be used to collect participants' demographic characteristics and basic information regarding their environmental attitudes. This form consists of 14 questions in total. In addition to demographic data such as participants' gender, grade level, age, and parents' educational background, the form includes items about participation in school activities related to nature and the environment, use of recycling bins at home, attitudes toward spending time in nature, knowledge levels about environmental and recycling issues, types of materials separated for recycling at home, frequency of time spent in nature, emotions felt when recycling is not practiced, family recycling habits, and interest in acquiring information about nature and environmental topics.
  The study data will be collected from selected middle schools affiliated with the Istanbul Directorate of National Education.

CONTACTS AND LOCATIONS:
Overall Officials: Merve KOLCU, PhD, Principal Investigator — merve.kolcu@sbu.edu.tr; Aydan YILMAZ, Msc, Study Chair — aydan.yilmaz@sbu.edu.tr
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No